CLINICAL TRIAL: NCT05463133
Title: Phase I/II Study Using Allogeneic Hematopoietic Stem Cell Transplantation for Chronic Granulomatous Disease With an Alemtuzumab, Busulfan and TBI-based Conditioning Regimen Combined With Cytokine (IL-6, +/- IFN-gamma) Antagonists
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation for Chronic Granulomatous Disease (CGD) With an Alemtuzumab, Busulfan and TBI-based Conditioning Regimen Combined With Cytokine (IL-6, +/- IFN-gamma) Antagonists
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000977; 000977-I
Record Dates: First submitted 2022-07-15; First posted 2022-07-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05-30

CONDITIONS: Chronic Granulomatous Disease
Keywords: HLA Matched Related Donor; Matched Unrelated Donor; The National Marrow Donor Program
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Sirolimus; Cyclophosphamide; Alemtuzumab; Busulfan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 / Group 1 Standard Risk (Active Comparator): Group 1 (Standard group) will receive tociluzumab at Day -10, Alemtuzumab on Day -9,-8,-7,-6,-5; Busulfan on Day -4, and -3, TBI, matched donor PBSC infusion, and Post transplant Cyclophosphamide.
  Interventions: Drug: Sirolimus; Drug: Cyclophosphamide; Drug: Alemtuzumab; Drug: Busulfan; Biological: Pheripheral blood stem cells; Drug: Tociluzumab; Drug: Total Body Irradiation
- Arm 2 / Group 2 High Risk. (Experimental): Group 2 (High risk group will receive tociluzumab at day -24, a repeat dose at day -19, Alemtuzumab at day -9,-8,-7,-6,-5; Busulfan at day -4 and -3, Emapalumab at Day -1, matched donor PBSC infusion, and post transplant cyclophosphamide at Day +3 and +4
  Interventions: Drug: Sirolimus; Drug: Cyclophosphamide; Drug: Alemtuzumab; Drug: Busulfan; Biological: Pheripheral blood stem cells; Drug: Emapalumab-Izsg; Drug: Tociluzumab

INTERVENTIONS:
Drug: Sirolimus — Post transplant drug - Immunosuppressant to prevent donor peripheral blood stem cell rejection and graft versus host disease. This is a well studied drug, and is not under an IND.
Drug: Cyclophosphamide — Post transplant drug - cyclophosphamide give to prevent graft versus host disease. This is a well studied drug and s not under an IND.
Drug: Alemtuzumab — Transplant Conditioning Drug - Monoclonal antibody that targets recipient and donor T-cells to prevent graft versus host disease. Not an IND. This is a well-studied drug, and is not under an IND.
Drug: Busulfan — Transplant Conditioning Drug - Chemotherapy to create space in the patient's bone marrow so that the donor peripheral blood stem cells can repopulate in the patient's bone marrow. This is a well studied drug, and is not under IND.
Biological: Pheripheral blood stem cells — Donor peripheral blood stem cells either matched unrelated donors or matched related relative to replace the patient's immune cells with functional immune cells. The peripheral blood stem cells are not regulated by the FDA.
Drug: Emapalumab-Izsg — Transplant conditioning drug for High Risk Group only - An interferon gamma blocking antibody used to prevent inflammation/engraftment syndrome post HSC transplant.
  Arms: Arm 2 / Group 2 High Risk.
Drug: Tociluzumab — Transplant Conditioning Drug - An interleukin-6 (IL-6) receptor antagonist used to decrease Chronic Granulomatous Disease (CGD) inflammation during the HSC transplant process.
Drug: Total Body Irradiation — Transplant Conditioning - Total Body Irradiation (300 cGy in fractionated doses) to create space n the subject's bone marrow so that the donor peripheral blood stem cells can repopulate in the subject's bone marrow.
  Arms: Arm 1 / Group 1 Standard Risk

SUMMARY:
Background:

Chronic granulomatous disease (CGD) affects the immune system. People with CGD are more likely to get infections. Drugs can help control infections, but these treatments can cause side effects including kidney failure and deafness. Stem cell transplants can cure CGD, but these don t always work.

Objective:

To find out if a different drug treatment can improve the success rates of stem cell transplants in people with CGD.

Eligibility:

People aged 4-65 years with CGD.

Design:

Participants will undergo screening. They will have a physical exam. They will have blood and urine tests and tests of their heart function and breathing. They will have imaging scans. They will have a bone marrow biopsy; a needle will be inserted into their hip to draw a sample of tissue from the bone.

A tube called a catheter will be placed into a vein in the participant s chest. This catheter will remain in place for the transplant and recovery period. Blood for tests can be drawn from the catheter, and medications and the stem cells can be administered through it.

Participants will be in the hospital for either 10 or 21 days to receive 3 or 4 drugs before the transplant. They will get 2 doses of total body radiation on the same day.

Participants will receive donor stem cells through the catheter. They will remain in the hospital for 6 weeks afterward.

Participants will visit the clinic 2 to 3 times per week for 3 months after discharge.

Follow-up visits will continue for 5 years.

DETAILED DESCRIPTION:
Chronic Granulomatous Disease (CGD) is an inherited disorder resulting from a failure to produce nicotinamide adenine dinucleotide phosphate (NADPH) oxidase, necessary for protection against a number of infectious organisms. Patients are subject to recurrent infections and inflammatory complications. The current management of these patients is limited to close surveillance for infections, administration of prophylactic antimicrobials, and rapid and aggressive treatment of suspected and documented infections with broad-spectrum antibiotics. Although often effective, these treatments can require long hospitalizations, impacting the overall quality of life significantly and leading to significant morbidity, such as renal failure and deafness. CGD patients have autoinflammation that may manifest as inflammatory bowel disease, hypoxic lung inflammation, and/or liver nodular regenerative hyperplasia with venopathy as examples.

Currently the only available cure for these disorders is bone marrow transplantation, which preferentially uses a human leukocyte antigen (HLA)-matched related sibling as the donor (allogeneic stem cell transplantation). However, as only 30% of participants in the general population have an HLA-matched related sibling, allogeneic related transplantation is often not an option, resulting in the need for matched unrelated donor (MUD) transplantation. The National Marrow Donor Program (NMDP) serves as both a national registry of volunteers who are willing to donate progenitor cells to eligible recipients as well as a repository of cord blood products. Despite continued improvement in the use of transplantation schemas- including the development of nonmyeloablative regimens-there remain significant morbidity and mortality associated with transplantation, in particular graft versus host disease (GvHD) and graft rejection. CGD with severe autoinflammation manifested as C-reactive protein (CRP) >=100 milligrams per milliliter (mg/mL) has been a significant risk factor for mortality due to severe engraftment syndrome, and thus patients with elevated CRPs have not been eligible for prior transplant protocols.

In addition, despite improving engraftment rates, there continues to be mixed chimerism and late graft loss in CGD participants despite a variety of conditioning regimens being used at various centers.

In our most recent protocol, we have continued to have a low incidence of graft versus host disease and improved engraftment, but still could see improvement in graft stability. Thus, in order to improve outcomes with participants with elevated CRPs as well as improve overall engraftment, we are building on our prior regimens by targeting the inflammatory cytokines that appear to be involved in graft failure and engraftment syndrome.

Participants with a CRP of less than 100 mg/mL will be pretreated with a dose of tocilizumab, an anti-IL6 monoclonal antibody. Participants with a CRP of greater than 100 mg/mL will be pretreated with 2 doses of tocilizumab as well as an inhibitor of interferon-gamma in order to decrease the inflammation that has been seen in these participants with engraftment. Otherwise, the conditioning regimen will be similar to maintain the low rates of GvHD that we have seen to date.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all the following criteria:

* Must have the ability to comprehend and a willingness to sign the informed consent. For pediatric patients, must have a parent/guardian who can sign consent if the donor is a minor; assent will be obtained from minors as appropriate.
* Must have confirmed diagnosis of CGD.
* Must have sufficient complications from underlying disease to warrant undergoing transplantation (either a history of or ongoing inflammation/CGD-related autoimmunity OR a CGD-related infection while on prophylaxis) OR have a Quartile 1 or 2 residual oxidase production level.
* Ages 4 years-65 years.
* HLA-matched family donor graft or an HLA-matched unrelated PBSC graft (10/10 or 9/10 mismatch) available.
* Must be human immunodeficiency virus (HIV) negative.
* When discharged from the hospital the participant must be able to stay within 1 hour s travel of the NIH for the first 3 months after transplantation.
* Must have a family member or other designated care provider to assist with care during the post-transplant period when the patient is in the outpatient setting.
* Must provide a durable power of attorney for health care decisions to an appropriate adult relative or guardian in accordance with NIH 200 'NIH Durable Power of Attorney for Health Care Decision Making.'
* Females of child-bearing potential must agree to consistently use one form of contraception from 1 month prior to study entry and for at least 1 year post transplant. Male participants must agree to consistently use contraception for 1 year post transplant. Acceptable forms of contraception are:

  * Contraceptive pills or patch, Norplant [Registered], Depo-Provera [Registered], or other FDA-approved contraceptive method.
  * Male partner has previously undergone a vasectomy.
  * Male participants will be advised to consistently use contraception throughout study participation and for 3 months post-transplant.
* Stated willingness to comply with all study procedures and is available for protocol visits for the duration of the study when possible.
* Patients who have a CRP of greater than 100 but otherwise meet inclusion criteria will be enrolled on the high-risk arm.

  * CRP will be assessed no more than 7 weeks and no less than 6 weeks prior to anticipated transplant to determine on which arm the patient will be treated.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Ejection fraction of less than 30% by echocardiography.
* Forced expiratory volume (FEV1%) of less than 35% and/or an adjusted diffusing capacity of lung of carbon monoxide (adj DLCO) of less than 30%.
* Transaminases >5x upper limit of normal based on the individual s clinical situation and at the discretion of the investigator.
* Psychiatric disorder or mental deficiency severe enough as to make compliance with the HSCT treatment unlikely, and/or to make regulatorily and legally effective informed consent impossible.
* Major anticipated illness or organ failure incompatible with survival from allogeneic peripheral blood stem cell (AlloPBSC) transplant.
* Pregnant or lactating.
* Uncontrolled seizure disorder per principal investigator (PI) discretion.
* Individuals older than 65 years are excluded. It is known from standard transplantation that these individuals have a higher risk of morbidity and mortality related to transplantation. Given the investigational nature of this protocol, the risk-benefit ratio is not warranted to include these individuals at this time.
* Active TB infection.
* Any condition or circumstance that the PI feels would create difficulty in maintaining compliance with the requirements of this protocol.
* Individuals who are not willing to submit their information as part of the alemtuzumab (Campath [Registered]) Distribution Program application or participants whom the Distribution Program committee has determined are not qualified to receive alemtuzumab.

NOTE: Alemtuzumab (Campath-1H) (intravenous [IV] formulation) is no longer distributed commercially. To receive product, the physician must contact the program for the patient. If the patient is not willing to consent to submit their info (demographics, contact information, and rationale for use) to the program such that we can obtain the drug, then we cannot proceed with conditioning; therefore no transplant will occur on this protocol. http://www.campath.com/

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 years post-transplant.
  Alive at 1 years post-transplant.

SECONDARY OUTCOMES:
To assess the infection rates in the setting of Alemtuzumab (Campath-1H) and post-transplant cyclophosphamide with the addition of an Il-6 antagonist and TNF inhibitor. | Day 100, 6 months, 1 and/or 2 years post BMT
  Any documented viral, bacterial, fungal, or parasitic infection.
To assess kinetics of engraftment | Day +14, +30, +60, +100, 6 month and 1 year post transplant
  Measurement of chimerism, lymphocyte phenotype (TBNK/SCID/TVB), and cytokine analysis laboratory values and research cytokine, alemtuzumab, and CXCL9 levels
Improve eligibility for allogeneic transplantation. | Eligibility determination for protocol enrollment
  Subject eligible to enroll in the protocol.
Engraftment without GvHD | Day 100, 6 months, and/or 1 year post BMT
  As defined by a >20% myeloid engraftment of donor neutrophils. Will be assess as event-free survival (EFS)
Decreased engraftment syndrome. | 30 days post transplant.
  Engraftment syndrome symptoms such as fever, erythrodermal rash, noncardiogenic pulmonary edema, hepatic dysfunction, renal insufficiency, weight gain and transient encephaopathy that is responsive to steroids and/or tocilizumab, and does not require ICU admission or lead to death.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The following date will be shared:@@@@@@All the individual participant data collected during the trial, after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data availability and the duration of the data availability are as follows: Transplant data shared with the following groups will be shared at the onset of the signing of the protocol and will be maintained in shared data bases with no end date. (BTRIS), Neutrophil Monitoring Laboratory (NML), The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people, NIH Intramural Institutional Review Board, The Center for Blood and Marrow Transplant Research, Study sponsor (NIAID), NHLBI s Data Safety and Monitoring Board, Blood and Inherited Disorder-Transplant and Cellular Therapy Program, Study monitors (NIAID/Office of Clinical Research Policy and Regulatory Operations NIAID/OCRPRO). Transplant data submitted for publication will be immediately available following publication with no end date.
Access Criteria: Individual deidentified participant data will be shared with: A public repository, (CIBMTR), as required by the Stem Cell Act 2005 through the Forms Net database system. An NIH-funded or approved public repository. Publications, Public presentations, Individual identified participant data will be shared, approved outside collaborators under appropriate agreements, such as the NMLab in Md. Identified data in (BTRIS). The following data will be shared: All the individual participant data collected during the trial, after deidentification. The following related documents will be available: Study Protocol, Statistical analysis plan, Analytic code. Data and the duration of the data availability are as follows: Transplant data shared with CIBMTR, BTRIS, and the NML will be shared at the onset of signing the protocol and will be maintained in shared databases with no end date. Transplant data submitted for publication will be immediately available following publication with no end date.

REFERENCES:
- [Background] Parta M, Kelly C, Kwatemaa N, Theobald N, Hilligoss D, Qin J, Kuhns DB, Zerbe C, Holland SM, Malech H, Kang EM. Allogeneic Reduced-Intensity Hematopoietic Stem Cell Transplantation for Chronic Granulomatous Disease: a Single-Center Prospective Trial. J Clin Immunol. 2017 Aug;37(6):548-558. doi: 10.1007/s10875-017-0422-6. Epub 2017 Jul 28. PMID 28752258
- [Background] Kadauke S, Myers RM, Li Y, Aplenc R, Baniewicz D, Barrett DM, Barz Leahy A, Callahan C, Dolan JG, Fitzgerald JC, Gladney W, Lacey SF, Liu H, Maude SL, McGuire R, Motley LS, Teachey DT, Wertheim GB, Wray L, DiNofia AM, Grupp SA. Risk-Adapted Preemptive Tocilizumab to Prevent Severe Cytokine Release Syndrome After CTL019 for Pediatric B-Cell Acute Lymphoblastic Leukemia: A Prospective Clinical Trial. J Clin Oncol. 2021 Mar 10;39(8):920-930. doi: 10.1200/JCO.20.02477. Epub 2021 Jan 8. PMID 33417474
- [Background] Chiesa R, Wang J, Blok HJ, Hazelaar S, Neven B, Moshous D, Schulz A, Hoenig M, Hauck F, Al Seraihy A, Gozdzik J, Ljungman P, Lindemans CA, Fernandes JF, Kalwak K, Strahm B, Schanz U, Sedlacek P, Sykora KW, Aksoylar S, Locatelli F, Stepensky P, Wynn R, Lum SH, Zecca M, Porta F, Taskinen M, Gibson B, Matthes S, Karakukcu M, Hauri-Hohl M, Veys P, Gennery AR, Lucchini G, Felber M, Albert MH, Balashov D, Lankester A, Gungor T, Slatter MA. Hematopoietic cell transplantation in chronic granulomatous disease: a study of 712 children and adults. Blood. 2020 Sep 3;136(10):1201-1211. doi: 10.1182/blood.2020005590. PMID 32614953
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000977-I.html